CLINICAL TRIAL: NCT00365456
Title: An Open Label, International, Multi Centre, Parallel Group, Phase III b, Randomised Trial, Investigating Lumbar Spine Bone Mineral Density (BMD) Changes in Postmenopausal Women With Primary Osteoporosis Initially Treated With 12 Months of Full Length Parathyroid Hormone (PTH 1-84) Followed by 12 Months of Treatment With Risedronate Followed by Either 12 Months Treatment With PTH (1-84) or Risedronate.
Brief Title: Sequential Treatment of Postmenopausal Women With Primary Osteoporosis (FP-001-IM)
Acronym: PEAK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP-001-IM; 2005-000730-20 (EudraCT Number); U1111-1132-3246 (Registry Identifier: WHO)
Record Dates: First submitted 2006-08-09; First posted 2006-08-17 (Estimated); Results first posted 2012-07-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Osteoporosis
Keywords: Lumbar Spine Bone Mineral Density (BMD)
MeSH Terms: conditions — Osteoporosis | interventions — Parathyroid Hormone; Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PTH (1-84) (Experimental)
  Interventions: Drug: Parathyroid Hormone (PTH)
- Risedronate (Active Comparator)
  Interventions: Drug: Risedronate

INTERVENTIONS:
Drug: Parathyroid Hormone (PTH) — Self-administered (100 μg in a volume of 71.4 μL) daily as a subcutaneous injection in the abdomen using the Preotact pen.
  Arms: PTH (1-84)
Drug: Risedronate — Orally once weekly as one 35 mg tablet.
  Arms: Risedronate

SUMMARY:
The objective is to show superior efficacy of PTH (1-84) over risedronate in treating osteoporotic women for 12 months after having previously been treated with PTH (1-84) for 12 months followed by 12 months treatment with risedronate.

ELIGIBILITY:
Inclusion Criteria:

Women above the age of 50 years with the diagnosis of postmenopausal primary osteoporosis may be enrolled in the trial if the following inclusion/exclusion criteria apply.

All inclusion criteria must be answered "yes" for a subject to be enrolled in the trial.

1. Has the subject given informed consent according to local requirements before any trial related activities? (A trial related activity is any procedure that would not have been performed during the routine management of the subject).
2. Is the subject above 50 years old?
3. Is the subject postmenopausal (more than 5 years) - in the judgement of the investigator?
4. Does the subject have primary osteoporosis with a lumbar spine T score < -3.0 SD (at lumbar spine L1-L4, with a minimum of two evaluable vertebrae)?
5. Does the subject have a life expectancy of >3 years?
6. Is the subject able to self-inject PTH (1-84), (or to have PTH (1-84) injection by a helper)?

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2006-07; Primary Completion 2011-01 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquaters
Locations (1):
- Roskilde, Denmark

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was divided into 3 consecutive open-label treatment phases of 12 months with randomisation after Trial Period II.
  From 407 enrolled patients in total, 2 patients were enrolled but were never exposed to trial treatment. Thus, 405 patients in total received trial treatment.
Pre-assignment Details: * Period I: total number of 405 patients were included and all received PTH(1-84) treatment for 1 year
  * Period II: of those 405 patients, 282 continued into the 2. year and all received risedronate
  * Period III: during the 3. year, the remaining 268 patients were randomised to either PTH(1-84) (=136 patients) or risedronate (=132 patients)
Period: Trial Period I (12 Months)
Arm/Group | PTH (1-84) | Risedronate
Started | 407 | 0
Completed | 282 | 0
Not Completed | 125 | 0
Not completed — Adverse Event | 84 | 0
Not completed — Non-compliance | 3 | 0
Not completed — Withdrawal by Subject | 27 | 0
Not completed — Other | 11 | 0
Period: Trial Period II (12 Months)
Arm/Group | PTH (1-84) | Risedronate
Started | 0 | 282
Completed | 0 | 268
Not Completed | 0 | 14
Not completed — Adverse Event | 0 | 6
Not completed — Non-compliance | 0 | 2
Not completed — Withdrawal by Subject | 0 | 5
Not completed — Other | 0 | 1
Period: Trial Period III (12 Months)
Arm/Group | PTH (1-84) | Risedronate
Started | 136 | 132
Completed | 118 | 127
Not Completed | 18 | 5
Not completed — Adverse Event | 13 | 3
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Other | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- PTH(1-84) or Risedronate: * PTH(1-84) received by 405 participants in Trial Period I
  * of those 405 participants, 282 received Risedronate in Trial Period II
  * of those 282 participants, 268 participant remained and 136 received PTH(1-84) and 132 received Risedronate in Trial Period III
Arm/Group | PTH(1-84) or Risedronate
Number analyzed (Participants) | 405
Age, Customized [Mean (Standard Deviation); unit: years]
  Trial Period I / PTH(1-84) | 64.6 (7.46)
  Trial Period II / Risedronate | 64.2 (7.43)
  Trial Period III / PTH(1-84) | 63.4 (6.94)
  Trial Period III / Risedronate | 64.7 (7.91)
Sex/Gender, Customized [Number; unit: participants]
  female | 405
Lumbar spine T-score [Mean (Standard Deviation); unit: score] — The T-score represents the lumbar spine bone mineral density as compared to a young normal reference mean (healthy 30-year-old woman). A score ≥ -1.0 is considered Normal, while a score between -1.0 and -2.5 is defined as Osteopenia and a score ≤ -2.5 is defined as Osteoporosis.
  score
    Trial Period I / PTH(1-84) | -3.61 (0.490)
    Trial Period II / Risedronate | -3.62 (0.472)
    Trial Period III / PTH(1-84) | -3.60 (0.427)
    Trial Period III / Risedronate | -3.63 (0.518)
Prevalent vertebral fractures [Number; unit: participants] — Number of patients with at least one vertebral fracture at baseline
  participants
    Trial Period I / PTH(1-84) | 105
    Trial Period II / Risedronate | 71
    Trial Period III / PTH(1-84) | 37
    Trial Period III / Risedronate | 29
Prevalent non-vertebral fragility fractures [Number; unit: participants]
  Trial Period I / PTH(1-84): hip fractures | 9
  Trial Period II / Risedronate: hip fractures | 5
  Trial Period III / PTH(1-84): hip fractures | 1
  Trial Period III / Risedronate: hip fractures | 3
  Trial Period I / PTH(1-84): wrist fractures | 78
  Trial Period II / Risedronate: wrist fractures | 50
  Trial Period III / PTH(1-84): wrist fractures | 22
  Trial Period III / Risedronate: wrist fractures | 25
  Trial Period I / PTH(1-84): others | 93
  Trial Period II / Risedronate: others | 59
  Trial Period III / PTH(1-84): others | 28
  Trial Period III / Risedronate: others | 27
Weight [Mean (Standard Deviation); unit: kg]
  Trial Period I / PTH(1-84) | 59.5 (9.39)
  Trial Period II / Risedronate | 59.7 (9.17)
  Trial Period III / PTH(1-84) | 59.6 (8.66)
  Trial Period III / Risedronate | 59.8 (9.57)
Height [Mean (Standard Deviation); unit: cm]
  Trial Period I / PTH(1-84) | 157.4 (6.40)
  Trial Period II / Risedronate | 157.5 (6.48)
  Trial Period III / PTH(1-84) | 157.6 (6.21)
  Trial Period III / Risedronate | 157.4 (6.86)
Serum Calcium [Mean (Standard Deviation); unit: mmol/L]
  Trial Period I / PTH(1-84) | 2.338 (0.1022)
  Trial Period II / Risedronate | 2.337 (0.0999)
  Trial Period III / PTH(1-84) | 2.337 (0.0961)
  Trial Period III / Risedronate | 2.339 (0.1041)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2]
  Trial Period I / PTH(1-84) | 24.06 (3.861)
  Trial Period II / Risedronate | 24.11 (3.788)
  Trial Period III / PTH(1-84) | 24.06 (3.618)
  Trial Period III / Risedronate | 24.21 (3.933)

OUTCOME MEASURES:

1. Primary Outcome: Change in Lumbar Spine BMD From Start of Trial Period III Until End of Trial Period III.
Description: BMD was measured by Dual X-ray Absorptiometry (DXA).
Time Frame: 12 months
Population: All randomized patients made the Full Analysis Set which was used for the primary and secondary analyses according to intention-to-treat principles. One participant excluded due to missing baseline data at trial period III entry, thus no data could be carried forward for this patient. Missing values imputed by Last Observation Carried Forward.
Measure: Least Squares Mean (Standard Error); unit: Percentage Change
Groups:
- PTH (1-84): Regimen 1 = PTH (1-84) → Risedronate → PTH (1-84)
- Risedronate: Regimen 2 = PTH (1-84) → Risedronate → Risedronate
Arm/Group | PTH (1-84) | Risedronate
Number analyzed (Participants) | 135 | 132
Percentage Change | 1.002 (1.0037) | 0.990 (1.0034)
Statistical Analysis 1: Comparison: PTH (1-84) vs Risedronate; An analysis of covariance (ANCOVA) model was used including treatment group, stratum and pooled centre as fixed effects and log (BMD at Baseline III (month 24)) as a covariate (log-normally distributed data assumed). Least square mean change from baseline III (month 24), 95% confidence interval and p-value for the treatment effect (PTH (1-84) vs. Risedronate) was calculated. Superiority was claimed if lower limit of the interval was above 1. Results were back-transformed from the log scale; Test type: Superiority or Other; p = 0.010, ANCOVA — No multiplicity correction of the significance level was performed as only one primary endpoint was planned; Estimation allowing for unequal variance in the two treatment groups and robust estimates for the standard errors were obtained; Mean Difference (Final Values) = 1.012, 95% CI 2-sided [1.003 to 1.021], Standard Error of Mean 1.0045

ADVERSE EVENTS:
Time Frame: Over three years of the trial duration.
Description: The safety analysis set (SAF) was defined as all subjects enrolled in Trial Period I who received at least one dose of the IMP.
  At each contact between the site and the subject (visit or phone) the subject was asked if she has experienced any health problems since the last contact.
Groups:
- PTH (1-84): Trial Period I SAEs and Trial Period III SAEs for subjects receiving PTH (1-84)
- Risedronate: Trial Period II SAEs and Trial Period III SAEs for subjects receiving risedronate
Arm/Group | PTH (1-84) | Risedronate
Serious Adverse Events (participants affected / at risk) | 33/405 | 32/282
Other Adverse Events (participants affected / at risk) | 365/405 | 95/282
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTH (1-84) (N=405) | Risedronate (N=282)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Eye disorder (Eye disorders) | 1 (1) | 0 (0)
Retinal detachment (Eye disorders) | 1 (1) | 0 (0)
Retinal vein thrombosis (Eye disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1)
Condition aggravated (General disorders) | 1 (1) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ulna fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Impacted fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 1 (1) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Mesothelioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 2 (2)
Nephrotic syndrome (Renal and urinary disorders) | 0 (0) | 1 (1)
Uterine polyp (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Bunion operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Medical device removal (Surgical and medical procedures) | 0 (0) | 1 (1)
Angiopathy (Vascular disorders) | 1 (1) | 0 (0)
Femoral arterial stenosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 1 (1)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PTH (1-84) (N=405) | Risedronate (N=282)
Vertigo (Ear and labyrinth disorders) | 24 (26) | 0 (0)
Nausea (Gastrointestinal disorders) | 98 (123) | 0 (0)
Asthenia (General disorders) | 23 (24) | 0 (0)
Urinary tract infection (Infections and infestations) | 23 (28) | 14 (16)
Influenza (Infections and infestations) | 0 (0) | 20 (24)
Hypercalcaemia (Metabolism and nutrition disorders) | 87 (105) | 17 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 31 (32) | 15 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 14 (16)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 15 (16)
Headache (Nervous system disorders) | 35 (40) | 0 (0)
Hypercalciuria (Renal and urinary disorders) | 121 (150) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After publication of the results or 24 months after Clinical Trial Report has been finalised, whichever comes first, Nycomed acknowledge the Investigator's rights to publish results from this trial. Any such scientific paper, presentation, communication, or other information concerning the investigation described in this protocol, must be submitted to Nycomed prior to submission for publication/presentation for review. Review comments will be given within a month from receipt of the manuscript.